CLINICAL TRIAL: NCT06715410
Title: CO2 Pilot Clinical Investigation
Brief Title: Carbon Dioxide Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21290936998
Record Dates: First submitted 2024-06-05; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Intubation; Tracheostomy; Laryngeal Mask

STUDY DESIGN:
Intervention Model Description: The purpose of this clinical study is to collect parameter raw data for development and to evaluate the operational and functional features as well as ease of use of the system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CO2 data collection (Other): To collect data from CO2
  Interventions: Device: CO2

INTERVENTIONS:
Device: CO2 — To collect CO2 data

SUMMARY:
The investigational device enables monitoring of EtCO2, FiCO2 and respiration rate values.

The purpose of this clinical study is to collect parameter raw data for development, evaluate the operational and functional features of the investigational device as well as ease of use of the system.

ELIGIBILITY:
Inclusion Criteria:

* Adults and pediatric patients that are endotracheally intubated, tracheostomized or have a laryngeal mask or similar
* Tolerate airway adapter dead space of 6.7 ml
* Are above 10 kg
* 2 years of age of older
* Able to provide written informed consent or have a LDR to provide written informed consent
* Are being cared for in hospital unit and are expected to remain in the unit for the duration of the study procedure

Exclusion Criteria:

* Are known to be pregnant
* Are breastfeeding
* Are suffering from infection(s) or immunocompromised patients that require isolation.
* PI or designee decision due to subject health condition

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Collection of data | From admission to discharge, maximum of 48 hours
  Raw parameter data will be collected from subjects in clinical settings.

SECONDARY OUTCOMES:
Evaluation of the performance and usability of CO2 measurement | From admission to discharge, maximum of 48 hours
  Research nurses will fill in questionnaires during the study

OTHER OUTCOMES:
To collect safety information | From admission to discharge, maximum of 48 hours
  Collection of type and number of AEs, SAEs, and device issues.

CONTACTS AND LOCATIONS:
Overall Officials: Tero Varpula, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Espoo, Uusimaa, Finland